CLINICAL TRIAL: NCT07184138
Title: Efficacy and Safety of Interleukin-23 Inhibitors (IL-23i) in the Treatment of Inflammatory Bowel Disease in China: A Multicenter, Single-Arm, Prospective, Observational Real-World Study
Brief Title: Real-World Study on the Safety and Effectiveness of IL-23 Inhibitors for Inflammatory Bowel Disease in China
Status: Not yet recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chao Kang, Clinical professor, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 20250913
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Inflamatory Bowel Disease (Crohn's and Ulcerative Colitis)
Keywords: IL23i; Crohn's disease; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult IBD Patients Treated With IL-23i: Adult patients diagnosed with ulcerative colitis (UC) or Crohn's disease (CD) in China who are initiating treatment with an interleukin-23 inhibitor (IL-23i) in a real-world clinical practice setting. Patients will be observed prospectively for treatment effectiveness and safety outcomes.
  Interventions: Drug: Interleukin-23 Inhibitors (IL-23i)

INTERVENTIONS:
Drug: Interleukin-23 Inhibitors (IL-23i) — Adult patients will receive treatment with an interleukin-23 inhibitor (IL-23i), including guselkumab or risankizumab, as prescribed in routine clinical practice in China. This observational study does not mandate dosing, administration schedule, or concomitant medications; treatments follow standard of care. Patients will be prospectively monitored for clinical effectiveness, endoscopic outcomes, and safety over 52 weeks.

SUMMARY:
Inflammatory bowel disease (IBD), including ulcerative colitis (UC) and Crohn's disease (CD), has shown greatly improved outcomes with biologic therapies. However, nearly half of patients still experience primary or secondary non-response to existing biologics. Interleukin-23 (IL-23), a member of the IL-12 cytokine family, plays a role in maintaining intestinal homeostasis but is also involved in the pathogenesis of IBD. IL-23 is a heterodimer composed of p19 and p40 subunits linked by a disulfide bond. Humanized monoclonal antibodies selectively targeting the IL-23 p19 subunit have emerged as promising therapies for IBD. Recently, selective IL-23p19 inhibitors-risankizumab (Risan) and mirikizumab-have been approved for the treatment of moderately to severely active CD and UC, respectively. In addition, these agents, along with guselkumab (Gus), are undergoing clinical trials for both CD and UC (guselkumab, gus, and mirikizumab for CD; guselkumab and risankizumab for UC). Guselkumab (Gus) and risankizumab (Risan), both targeting the IL-23 p19 subunit, have been approved in China for the treatment of CD, with guselkumab also approved for UC. However, data on the efficacy and safety of IL-23 inhibitors (IL-23i) in Chinese UC and CD patients remain limited, and evidence in Chinese IBD populations is lacking. This is a multicenter, single-arm, prospective, observational real-world study designed to evaluate the efficacy and safety of IL-23i in adult UC and CD patients in routine clinical practice in China.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older, any gender. Formally diagnosed with ulcerative colitis (UC) or Crohn's disease (CD). Determined by the treating physician to require initiation of IL-23 inhibitor (IL-23i) therapy for the first time.

Exclusion Criteria:

Currently enrolled in or planning to participate in any other interventional clinical study.

Contraindications to IL-23i treatment as specified in the drug label. Considered by the investigator to be unsuitable for participation in the study for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients in China diagnosed with ulcerative colitis (UC) or Crohn's disease (CD) who are initiating treatment with an interleukin-23 inhibitor (IL-23i) for the first time in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
clinical remission rate | Week 52
  To evaluate the effectiveness of IL-23 inhibitors (IL-23i) in real-world adult patients with ulcerative colitis (UC) or Crohn's disease (CD) by assessing clinical remission at Week 52

SECONDARY OUTCOMES:
clinical response rate | week 52
  To assess the real-world effectiveness of IL-23i in adult UC or CD patients by evaluating clinical response at Week 52
endoscopic remission rate | Week 52
  To evaluate endoscopic remission at Week 52 in adult UC or CD patients receiving IL-23i in routine clinical practice
endoscopic response rate | week 52
  To evaluate endoscopic response at Week 52 in adult UC or CD patients receiving IL-23i in routine clinical practice
Incidence of adverse events (AEs) and serious adverse events (SAEs) through Week 52 | Week 52
  To assess the safety of IL-23i in adult UC and CD patients by recording all adverse events (AEs) and serious adverse events (SAEs) occurring during the 52-week observation period

IPD SHARING:
Plan to Share IPD: No